CLINICAL TRIAL: NCT00940420
Title: Safety and Tolerability of Ribavirin (Ro 20-9963) in Combination With Peginterferon Alfa in Patients With Chronic Hepatitis C
Brief Title: A Study of Combination Treatment With Pegasys (Peginterferon Alfa) and Copegus (Ribavirin)in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML16837
Record Dates: First submitted 2009-07-06; First posted 2009-07-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (2):
- A (Experimental)
  Interventions: Drug: Copegus (ribavirin); Drug: peginterferon alfa-2a [Pegasys]
- B (Experimental)
  Interventions: Drug: Copegus (ribavirin); Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Copegus (ribavirin) — 800 - 1200 mg po daily for 24 weeks
  Arms: A
Drug: Copegus (ribavirin) — 800 - 1200 mg po daily for 48 weeks
  Arms: B
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc once weekly for 24 weeks
  Arms: A
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc once weekly for 48 weeks
  Arms: B

SUMMARY:
This 2 arm open-label study will assess the safety and tolerability of combination treatment with Peginterferon alfa (Pegasys) and Ribavirin (Copegus) in patients with chronic hepatitis C. Patients will be assigned to receive Peginterferon alfa (Pegasys) 180 mcg sc once a week and Ribavirin (Copegus) 800 - 1200 mg po daily for either 24 or 48 weeks. Allocation to the treatment arms is to the discretion of the investigator (mainly according to genotype). Adverse events will be monitored throughout the study and hematologic parameters every 2 weeks and twice during the 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/= 18 years of age
* serologic evidence of chronic hepatitis C infection
* compensated liver disease
* negative pregnancy test and in both males and females use of 2 forms of contraception during study and 6 months after treatment

Exclusion Criteria:

* history or other evidence of a medical condition associated with chronic liver disease other than HCV
* hepatitis A, hepatitis B or HIV infection
* hepatocellular carcinoma
* severe concomitant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2695 (Actual)
Dates: Start 2002-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
safety and tolerability with regard to clinical AEs and laboratory parameters | assessed every 2 weeks throughout study and after 8 weeks follow-up

SECONDARY OUTCOMES:
safety with regard to hematological parameters | assessed every 2 weeks throughout study and after 8 and 24 weeks of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Israel (17):
  - Afula
  - Ashkelon
  - Bat Yam
  - Beersheba
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Safed
  - Tel Aviv
  - Ẕerifin